CLINICAL TRIAL: NCT00318318
Title: Beneficial Effects of Oral Premarin Estrogen Replacement Therapy Assessed by Human Genome Array
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. G. Reid, Lawson Health Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R-06-710; GR12198E
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Healthy; Estrogen Replacement Therapy
Keywords: Premarin,; HRT,; RNA,; Gene Expression.; Postmenopausal Women
MeSH Terms: interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Premarin

SUMMARY:
The purpose of this study is to assess the immunological status of patients using Premarin. Premarin use is associated with an enhanced immune status, and possibly even some anti-cancer effect. The researchers will compare the use of Premarin with those not using hormone replacement therapy (HRT) to track the effects of Premarin in reducing the risk of infection and swelling.

DETAILED DESCRIPTION:
In recent times, adverse publicity has affected the sales of hormone replacement therapies and the perception of women as to whether or not HRTs should be taken. While a number of brands are available, those from Wyeth are the market leaders. Previous studies by our group have shown an advantage of Premarin, a natural conjugated equine estrogen, in fostering recovery of the Lactobacillus flora in the vagina. These organisms have been shown to help protect the host from urinary and vaginal infections. In the present proposal, we aim to further examine the beneficial effects of Premarin through the use of a human genome array technology.

New microarrays allow measurements to be made of 38,000 or more gene expressions on a single sample. We have recently used an Affymetrix array to examine up and down regulation of vaginal genes from a healthy premenopausal woman before and after administration of a probiotic. Somewhat to our surprise, we noted that over 9,000 genes were expressed and major down regulation occurred in cancer and other genes such as inflammatory cytokines. This was especially interesting as it showed that vaginal treatment could influence genes associated with, for example, the intestine. The array provided data or relevance to estrogen replacement therapy, namely the ability to detect and examine changes in estrogen associated factors.

In short, this system can examine changes to inflammation and host defenses. Based upon the findings of Raz and others (1993), it is likely that Premarin down regulates inflammation, either directly or via an alteration of the vaginal environment resulting in restoration of lactobacilli. Another benefit of the restoration of lactobacilli is that these organisms have anti-cancer properties.

The increased prevalence after menopause of urogenital (bladder and vaginal) infections and complications can be counteracted to some extent by restoration of the normal vaginal microbiota. These infections are extremely common, and treatment with antibiotics and antifungals is compromised by rapid rises in drug resistance (up to 30% for fluoroquinolones in some countries and a doubling of resistance to trimethoprim-sulfamethoxazole). BV has been associated with increased risk of preterm labour (McGregor et al. 1993; Hay et al. 1994; Chaim et al. 1997) and sexually transmitted diseases including HIV, herpes simplex virus, gonorrhea and Chlamydia (Sewankambo et al. 1997; Taha et al. 1998; Olinger et al. 1999; Wiesenfeld et al. 2003; Cherpes et al. 2003). Notably, 35-50% of patients and around 50% of UTI patients suffer a recurrence of infection within 3 months. Post-menopausal women have low levels of lactobacilli and high numbers of pathogens, while 100% of those receiving Premarin are colonized by lactobacilli (Burton et al. 2003; Devillard et al. 2004; Heinemann & Reid, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Women taking oral Premarin at least for the last month with no urogenital anatomical abnormalities.
* Women not taking HRT for at least one month with no urogenital anatomical abnormalities (controls).

Exclusion Criteria:

* Males.
* Subjects who are not menopausal.
* Less than 35 years of age.
* Subjects with recurrent sexually transmitted disease.
* Subjects with abnormal renal function (serum creatinine >110umol/l, upper limit 90umol/l) or pyelonephritis.
* Subjects receiving prednisone or immunosuppressive drugs,
* Subjects who need to be treated for any urogenital infection or with any antimicrobial therapy.
* Personal history of known or suspected estrogen-dependent neoplasia such as breast or endometrial cancer.
* Undiagnosed abnormal vaginal bleeding.
* Active hepatic dysfunction or disease, especially of the obstructive type.
* Active thrombophlebitis, thrombosis or thromboembolic disorders.
* Endometrial hyperplasia.
* Subjects on anticoagulants, antidiabetic and antihypertensive agents

Ages: 35 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Human genome array

SECONDARY OUTCOMES:
Denaturing gradient gel electrophoresis

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, MBA, Principal Investigator — Lawson Health Research Institute and The University of Western Ontario
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

REFERENCES:
- [Background] McGregor JA, French JI, Seo K. Premature rupture of membranes and bacterial vaginosis. Am J Obstet Gynecol. 1993 Aug;169(2 Pt 2):463-6. doi: 10.1016/0002-9378(93)90342-g. PMID 8357046
- [Background] Hay PE, Lamont RF, Taylor-Robinson D, Morgan DJ, Ison C, Pearson J. Abnormal bacterial colonisation of the genital tract and subsequent preterm delivery and late miscarriage. BMJ. 1994 Jan 29;308(6924):295-8. doi: 10.1136/bmj.308.6924.295. PMID 8124116
- [Background] Chaim W, Mazor M, Leiberman JR. The relationship between bacterial vaginosis and preterm birth. A review. Arch Gynecol Obstet. 1997;259(2):51-8. doi: 10.1007/BF02505309. PMID 9059744
- [Background] Sewankambo N, Gray RH, Wawer MJ, Paxton L, McNaim D, Wabwire-Mangen F, Serwadda D, Li C, Kiwanuka N, Hillier SL, Rabe L, Gaydos CA, Quinn TC, Konde-Lule J. HIV-1 infection associated with abnormal vaginal flora morphology and bacterial vaginosis. Lancet. 1997 Aug 23;350(9077):546-50. doi: 10.1016/s0140-6736(97)01063-5. PMID 9284776
- [Background] Taha TE, Gray RH, Kumwenda NI, Hoover DR, Mtimavalye LA, Liomba GN, Chiphangwi JD, Dallabetta GA, Miotti PG. HIV infection and disturbances of vaginal flora during pregnancy. J Acquir Immune Defic Syndr Hum Retrovirol. 1999 Jan 1;20(1):52-9. doi: 10.1097/00042560-199901010-00008. PMID 9928730
- [Background] Kalman S, Mitchell W, Marathe R, Lammel C, Fan J, Hyman RW, Olinger L, Grimwood J, Davis RW, Stephens RS. Comparative genomes of Chlamydia pneumoniae and C. trachomatis. Nat Genet. 1999 Apr;21(4):385-9. doi: 10.1038/7716. PMID 10192388
- [Background] Patrick DM, Dawar M, Cook DA, Krajden M, Ng HC, Rekart ML. Antenatal seroprevalence of herpes simplex virus type 2 (HSV-2) in Canadian women: HSV-2 prevalence increases throughout the reproductive years. Sex Transm Dis. 2001 Jul;28(7):424-8. doi: 10.1097/00007435-200107000-00011. PMID 11460028
- [Background] Wiesenfeld HC, Hillier SL, Krohn MA, Landers DV, Sweet RL. Bacterial vaginosis is a strong predictor of Neisseria gonorrhoeae and Chlamydia trachomatis infection. Clin Infect Dis. 2003 Mar 1;36(5):663-8. doi: 10.1086/367658. Epub 2003 Feb 7. PMID 12594649
- [Background] Cherpes TL, Meyn LA, Krohn MA, Hillier SL. Risk factors for infection with herpes simplex virus type 2: role of smoking, douching, uncircumcised males, and vaginal flora. Sex Transm Dis. 2003 May;30(5):405-10. doi: 10.1097/00007435-200305000-00006. PMID 12916131
- [Background] Devillard E, Burton JP, Hammond JA, Lam D, Reid G. Novel insight into the vaginal microflora in postmenopausal women under hormone replacement therapy as analyzed by PCR-denaturing gradient gel electrophoresis. Eur J Obstet Gynecol Reprod Biol. 2004 Nov 10;117(1):76-81. doi: 10.1016/j.ejogrb.2004.02.001. PMID 15474249
- [Background] Burton JP, Reid G. Evaluation of the bacterial vaginal flora of 20 postmenopausal women by direct (Nugent score) and molecular (polymerase chain reaction and denaturing gradient gel electrophoresis) techniques. J Infect Dis. 2002 Dec 15;186(12):1770-80. doi: 10.1086/345761. Epub 2002 Nov 22. PMID 12447763
- [Background] Heinemann C, Reid G. Vaginal microbial diversity among postmenopausal women with and without hormone replacement therapy. Can J Microbiol. 2005 Sep;51(9):777-81. doi: 10.1139/w05-070. PMID 16391657
- [Background] Notterman DA, Alon U, Sierk AJ, Levine AJ. Transcriptional gene expression profiles of colorectal adenoma, adenocarcinoma, and normal tissue examined by oligonucleotide arrays. Cancer Res. 2001 Apr 1;61(7):3124-30. PMID 11306497
- [Background] Habis AH, Vernon SD, Lee DR, Verma M, Unger ER. Molecular quality of exfoliated cervical cells: implications for molecular epidemiology and biomarker discovery. Cancer Epidemiol Biomarkers Prev. 2004 Mar;13(3):492-6. PMID 15006929
- [Background] Chen B, Wen Y, Zhang Z, Guo Y, Warrington JA, Polan ML. Microarray analysis of differentially expressed genes in vaginal tissues from women with stress urinary incontinence compared with asymptomatic women. Hum Reprod. 2006 Jan;21(1):22-9. doi: 10.1093/humrep/dei276. Epub 2005 Aug 26. PMID 16126751
- [Derived] Dahn A, Saunders S, Hammond JA, Carter D, Kirjavainen P, Anukam K, Reid G. Effect of bacterial vaginosis, Lactobacillus and Premarin estrogen replacement therapy on vaginal gene expression changes. Microbes Infect. 2008 May;10(6):620-7. doi: 10.1016/j.micinf.2008.02.007. Epub 2008 Feb 21. PMID 18485781